CLINICAL TRIAL: NCT04270292
Title: Arteriovenous Fistula Cannulation Methods and Dialysis Adequacy: A Cross-sectional Study From Turkey
Brief Title: Arteriovenous Fistula Cannulation Practices and Dialysis Adequacy
Status: Completed | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Assistant Professor, Istanbul Demiroglu Bilim University
Other Study IDs: P0139R00
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2020-05-22 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Arteriovenous Fistula; Hemodialysis; Dialysis Adequacy
Keywords: Arteriovenous fistula; Antegrade direction; Dialysis adequacy; Nursing care; Cannulation practices
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arteriovenous fistulae are preferred among methods of providing blood access for hemodialysis. For each hemodialysis treatment, the fistula is cannulated usually with two needles. One, the arterial needle, allows the blood to be withdrawn from the patient into the dialysis circuit and then it is returned by the second or venous needle. The success of arteriovenous fistula cannulation is dependent on many variables and these are affect the dialysis adequacy.

DETAILED DESCRIPTION:
As hemodialysis prescriptions are usually three times weekly (4 to 8 h), a fistula or graft for hemodialysis will be punctured twice each dialysis treatment or at least 312 times per year. To allow healing of the tissues damaged during each cannulation, optimal cannulation practice is required by rotation of the needle insertion sites each dialysis treatment. Vascular access (VA) has been justly described as both the lifeline and the Achilles' heel of hemodialysis therapy, making blood purification itself possible while simultaneously often constituting a limiting factor in treatment adequacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older years of age
* Have arteriovenous fistula
* Being on hemodialysis therapy for 4 hours a day on 3 days per week for at least 6 months
* Volunteering to participate in the study
* Have not communication problem

Exclusion Criteria:

* Younger than 18 years old
* Not volunteering to participate in the study
* Have communication problem
* Being on shorter hemodialysis therapy for 4 hours a day on 3 days per week for at least 6 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Being on hemodialysis therapy for 4 hours a day on 3 days per week for at least 6 months and 18 and older years of age who has arteriovenous fistula
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Asst. Prof., Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coventry LL, Hosking JM, Chan DT, Coral E, Lim WH, Towell-Barnard A, Twigg DE, Rickard CM. Variables associated with successful vascular access cannulation in hemodialysis patients: a prospective cohort study. BMC Nephrol. 2019 May 31;20(1):197. doi: 10.1186/s12882-019-1373-3. PMID 31151432
- [Background] Elias M, Nnang-Obada E, Charpentier B, Durrbach A, Beaudreuil S. Impact of arteriovenous fistula cannulation on the quality of dialysis. Hemodial Int. 2018 Jan;22(1):45-49. doi: 10.1111/hdi.12539. Epub 2017 Mar 6. PMID 28263032
- [Background] Gauly A, Parisotto MT, Skinder A, Schoder V, Furlan A, Schuh E, Marcelli D. Vascular access cannulation in hemodialysis patients - a survey of current practice and its relation to dialysis dose. J Vasc Access. 2011 Oct-Dec;12(4):358-64. doi: 10.5301/JVA.2011.8413. PMID 21688239
- [Derived] Ozen N, Aydin Sayilan A, Sayilan S, Mut D, Akin EB, Ecder ST. Relationship between arteriovenous fistula cannulation practices and dialysis adequacy: A prospective, multicenter study. J Ren Care. 2022 Mar;48(1):41-48. doi: 10.1111/jorc.12365. Epub 2021 Jan 25. PMID 33492745

RESULTS

PARTICIPANT FLOW:
Groups:
- Arteriovenous Fistula Cannulation Group: The cannulation practices' of patients was asked to the nurses and patients.
Period: Overall Study
Arm/Group | Arteriovenous Fistula Cannulation Group
Started | 164
Completed | 164
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arteriovenous Fistula Cannulation Group
Number analyzed (Participants) | 164
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [51 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Fistula Needle Direction
Description: The hemodialysis nurse who cannulate the patient's fistula fill the data form. There is two options about fistula direction as antegrade or retrograde.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arteriovenous Fistula Cannulation Group
Number analyzed (Participants) | 164
Participants
  Antegrade direction | 72
  Retrograde direction | 92

2. Primary Outcome: Number of Cannulation Method
Description: The hemodialysis nurse who cannulate the patient's fistula fill the data form. There is three options about cannulation method as puncture, buttonhole, and rope ladder methods.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arteriovenous Fistula Cannulation Group
Number analyzed (Participants) | 164
Participants
  Area puncture | 87
  Rope ladder | 54
  Buttunhole | 23

3. Primary Outcome: Number of Fistula Needle Rotated
Description: The researchers look to the fistula needle while it inserts to the fistula. There is two options as needle rotation is yes or no.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arteriovenous Fistula Cannulation Group
Number analyzed (Participants) | 164
Participants
  Yes | 104
  No | 60

4. Primary Outcome: Number of Arterial and Venous Needle Been on the Same Line
Description: The researchers look to the arterial and venous line whether they are the same venous line.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arteriovenous Fistula Cannulation Group
Number analyzed (Participants) | 164
Participants
  Yes | 25
  No | 139

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Arteriovenous Fistula Cannulation Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04270292/Prot_SAP_000.pdf